CLINICAL TRIAL: NCT03110666
Title: Treatment for Knee Osteoarthritis With Injections of Autologous Concentrated Bone Marrow Aspirate at the Bone-cartilage Interface Via Percutaneous. Pilot Study
Brief Title: Treatment for Knee Osteoarthritis With Injections of BMC at the Bone-cartilage Interface. Pilot Study
Acronym: IOC-target
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IOC-target
Record Dates: First submitted 2017-03-30; First posted 2017-04-12 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis ,; bone marrow aspirate; injections
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: autologous concentrated bone marrow aspirate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous concentrated bone marrow aspirate (Experimental): autologous concentrated bone marrow aspirate obtained from the BioCUE Concentration System
  Interventions: Biological: Injection of autologous concentrated bone marrow aspirate

INTERVENTIONS:
Biological: Injection of autologous concentrated bone marrow aspirate — Percutaneous injections at the bone-cartilage interface (distal femur and proximal tibia)

SUMMARY:
This pilot study will evaluate the clinica! and radiological results of a treatment for knee osteoarthritis with injections of autologous concentrated bone marrow aspirate at the bone-cartilage interface via percutaneous.

DETAILED DESCRIPTION:
This pilot study (N=30) patients will evaluate the clinica! and radiological results of a treatment for knee osteoarthritis with injections of bone marrow concentrate (BMC),obtained from the Bone Marrow Aspirate Concentration System (BioCUE) at the bone-cartilage interface via percutaneous injections. The PerFuse system will also be evaluated to determine if it can be used to deliver the BMC to the osseous sites. Follow-up is 1, 3, 6, 12, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* age ranging from 40 to 75
* Osteoarthritis of the medial or lateral compartment (2-3-4 grade according to the Kellgren-Lawrence score);
* Failure after at least 6 months of conservative treatment (drug therapy with NSAIDs,hyaluronic acid,platelet-rich plasma and corticosteroids injections);
* Signature of informed consent.

Exclusion Criteria:

* Patients with trauma in the 6 months prior to the intervention;
* Patients with malignancies;
* Patients with rheumatic diseases;
* Patients with diabetes;
* Patients suffering from metabolic disorders of the thyroid;
* Patients being abuse of alcohol, drugs or medications;
* Body Mass Index> 35;

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-11-14 (Actual); Primary Completion 2018-11-25 (Actual); Study Completion 2022-05 (Actual)

PRIMARY OUTCOMES:
improvement of the International Knee Documentation Committee (IKDC) subjective score | Time Frame: 1,3,6, 12, 24 months evaluation
  (International Knee Documentation Committee)

SECONDARY OUTCOMES:
improvement of the Knee Injury and osteoarthritis Outcome Score (KOOS) | Time Frame: 1,3,6, 12, 24 months evaluation
  (Knee Injury and osteoarthritis Outcome Score)
evaluation of WORMS score for MRI | Time Frame: 6, 12, 24 months evaluation
  MRI score

CONTACTS AND LOCATIONS:
Overall Officials: Elizaveta Kon, MD, Study Director — Rizzoli Orthopedic Institute
Locations (1):
- Rizzoli Orthopaedic Institute, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No